CLINICAL TRIAL: NCT05008341
Title: A Phase 4, Open-Label, Single-Dose Study to Evaluate Sunosi® (Solriamfetol) Pharmacokinetics in Breast Milk and Plasma of Healthy Postpartum Women Following Oral Administration of Sunosi®
Brief Title: Evaluate Sunosi® PK in Breast Milk and Plasma of Healthy Postpartum Women Following Single Dose Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZP110-401
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Narcolepsy; Obstructive Sleep Apnea; Excessive Daytime Somnolence; Excessive Sleepiness; Postpartum
Keywords: Sunosi; Solriamfetol; Healthy Postpartum Women; Breast Milk; Plasma
MeSH Terms: conditions — Narcolepsy; Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — solriamfetol; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Solriamfetol (Experimental): Participants will receive a single oral dose of solriamfetol 150 mg with 240 mL water at 0 hour on the morning of Day 1, 2 hours after completion of a light breakfast.
  Interventions: Drug: Solriamfetol 150 mg Oral Tablet

INTERVENTIONS:
Drug: Solriamfetol 150 mg Oral Tablet — Single-dose 150 mg tablet orally administered.
  Other Names: Sunosi®

SUMMARY:
The purpose of study JZP110-401 is to evaluate solriamfetol pharmacokinetics (PK) in the breast milk and plasma of healthy postpartum women following the administration of the drug. The study also aims to estimate the potential daily solriamfetol dose received by the infant from the breast milk of the nursing mother. The safety and tolerability of single oral doses of solriamfetol will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult female 18 to 50 years of age, inclusive, at the time of consent.
2. Weigh at least 50 kg, and have a body mass index within 18 to 35 kg/m2 inclusive.
3. Between 10 days and 52 weeks postpartum, inclusive, after delivery of a normal, healthy infant by the time of dosing, and actively lactating from both breasts.
4. If breastfeeding, agree to withhold breastfeeding their infant(s) from approximately 2 hours before dosing to approximately 72 hours after dosing and resume breastfeeding after completion of study Day 4 procedures OR have made a decision to wean their infant(s) before enrollment in the study.
5. Agree not to use nicotine-containing products including tobacco (cigarettes, cigars, chewing tobacco, snuff), e-cigarettes, and nicotine lozenge/gum/patch within 3 days prior to check-in on Day -1, and for the duration of the study.
6. Have used a medically acceptable method of contraception for at least the 2 months prior to dosing on Day 1, and consent to use a medically acceptable method of contraception throughout the entire study period and for 30 days after the study is completed.
7. Agree to comply with study-specified diet while in the study.
8. Able to understand and comply with study requirements.
9. Ensure that their breastfed infant(s) is able to feed from a bottle before study participation begins.
10. Agree to ensure nutrition is available for their infant(s) through stored breast milk, or alternative nutritional sources as necessary, for the duration of the study.

Exclusion Criteria:

1. Are pregnant.
2. History of any illness, physical finding, laboratory examination or electrocardiogram (ECG) finding that, in the opinion of the investigator, might confound the results or conduct of the study or pose a risk to the participant.
3. History or presence of gastrointestinal, hepatic, or renal disease or any other condition that may interfere with absorption, distribution, metabolism, or excretion of drugs.
4. Estimated creatinine clearance of < 90 mL/min.
5. History of breast implants, breast augmentation, or breast reduction surgery.
6. Presence of mastitis or other condition that would prevent the collection of milk from one or both breasts.
7. Presence of active suicidal ideation as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS).
8. History or presence of any clinically significant cardiovascular conditions.
9. Resting supine systolic blood pressure > 140 mmHg or < 90 mmHg or supine diastolic blood pressure > 90 mmHg or < 50 mmHg at the Screening Visit or at predose on Day 1. Blood pressure measurement may be repeated once at the discretion of the investigator.
10. Resting supine pulse rate of < 45 beats per minute (bpm) or >100 bpm at the Screening Visit or at predose on Day 1. Pulse rate measurement may be repeated once at the discretion of the investigator.
11. Unwilling to refrain from, or anticipates the use of, any medication, including prescription (with the exception of contraceptive agents) and non-prescription drugs (with the exception of acetaminophen no more than 2600 mg a day and ibuprofen no more than 1200 mg a day), antacids, vitamin supplements, or herbal remedies, beginning 14 days or 5 half-lives (whichever is longer) prior to Day 1 through the completion of breast milk collection and blood sampling.
12. Use of a monoamine oxidase inhibitor within 14 days prior to Day 1 through the completion of breast milk collection and blood sampling.
13. Unwilling to abstain from alcohol or caffeine/xanthine-containing products, including coffee, tea, chocolate, and cola, within 48 hours prior to Day 1 through the completion of breast milk collection and blood sampling.
14. Self-reported routine consumption of more than 600 mg of caffeine per day.
15. Positive breath alcohol or urine drug screen (including cannabinoids) at screening or at any point throughout the duration of the study.
16. Current or past (within the past 2 years) diagnosis of a moderate or severe substance use disorder according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria.
17. Current or history (within the past 2 years) of seeking treatment for a substance related disorder.
18. History or presence of phenylketonuria or a hypersensitivity or idiosyncratic reaction to phenylalanine-derived products, or any excipient in the formulated drug product.
19. Has participated in another clinical trial of an investigational drug or medical device within 30 days or five half-lives (whichever is longer) prior to Day 1.
20. Any other condition that would cause a risk to the participant if they participate in the trial, or to the ability of the participant to complete the study, based on the judgement of the investigator.
21. Employee of the study unit or Jazz Pharmaceuticals, anyone involved in the conduct of the trial, and first- and second-degree family member of anyone involved in the conduct of the trial.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) of Solriamfetol in Breast Milk and Plasma | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  The observed maximum breast milk and plasma concentrations (Cmax) of solriamfetol after administration.
Time to Reach Maximum Concentration (Cmax) (Tmax) in Breast Milk and Plasma | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  The time to reach the maximum breast milk and plasma concentrations (Tmax) of solriamfetol after administration.
Area Under the Concentration-Time Curve From Time 0 to the Time t of the Last Quantifiable Concentration (AUC 0-t) in Breast Milk and Plasma | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  The area under the plot of breast milk and plasma concentrations of solriamfetol against time after drug administration from predose (time 0) to Time t of the Last Quantifiable Concentration.
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC 0-inf) in Breast Milk and Plasma | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  The area under the plot of breast milk and plasma concentrations of solriamfetol against time after drug administration from predose (time 0) to Infinity.
Apparent Elimination Half-Life (t^1/2) of Solriamfetol in Breast Milk and Plasma | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  The half-life or the period of time required for the concentration of solriamfetol in breast milk and plasma to be reduced to one-half of the administered amount.
Apparent Oral Clearance (CL/F) of Solriamfetol | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  Apparent oral clearance (CL/F) of solriamfetol in plasma.
Apparent Volume of Distribution (Vd/F) of Solriamfetol | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  Apparent volume of distribution (Vd/F) of solriamfetol in plasma.
Milk:Plasma Ratio | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  Area Under the concentration-time curve (AUC) in breast milk divided by AUC in plasma.
Amount Excreted in Breast Milk Over 72 Hours (Amilk) | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  The amount of solriamfetol excreted in breast milk samples over 72 hours.
Daily Infant Dose | Predose, 1, 1.5, 3, 6, 8.5, 10, 13, 15, 21, 24, 28, 36, 44, and 72 hours post-dose.
  Daily solriamfetol dose that may be received by the infant through breastfeeding.
Relative Infant Dose | Up to 24 hours post-dose.
  The percentage of the weight-adjusted maternal solriamfetol dose excreted in breast milk over 24 hours.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Predose (-2 to 0 hours) up to Days 9-11 post-dose.
  A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) that either began after first study drug dose or worsened after dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- M3-Wake Research, Inc., Raleigh, North Carolina, United States

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com